CLINICAL TRIAL: NCT05371951
Title: A Pilot Evaluation of the Effect of the Erchonia® HLS™ on Individuals With Erectile Dysfunction
Brief Title: Effect of Erchonia Laser on Erectile Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in study subject recruitment
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-ED
Record Dates: First submitted 2022-05-04; First posted 2022-05-12 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Erchonia HLS (Experimental): 635 nanometers (nm) laser application
  Interventions: Device: Erchonia HLS

INTERVENTIONS:
Device: Erchonia HLS — 84 procedure administrations with the Erchonia® HLS™ administered by the subject at home: twice daily procedure administrations for 6 weeks.

SUMMARY:
This study is to see if applying low-level laser light can provide improvement in erectile dysfunction

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine the effectiveness of the Erchonia® HLS™, manufactured by Erchonia Corporation (the Company), in providing improvement in erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Male between 40 and 80 years old
* Known or suspected vasculogenic ED based on clinical history
* In an active sexual relationship with a minimum of 2 sexual attempts per month for at least one month prior to enrollment
* Suffering from ED for at least 6 months
* Testosterone level between 300 - 1000ng/dL within one month prior to enrollment
* Hgb A1C less than or equal to 8% within one month prior to enrollment
* Total IIEF-EF scores between 8-25
* EHS score greater than or equal to

Exclusion Criteria:

* ED due to radical prostatectomy, prior pelvic surgery, or radiation therapy to the pelvis within 12 months prior to enrollment
* Men with known neurogenic or psychogenic ED
* Anatomic malformations of the penis including Peyronie's disease
* Testosterone greater than 300ng/dL or 1000ng/dL
* Hgb A1C greater than 8%
* International Normalized Ratio greater than 2.5, and men on any blood thinners other than 81mg aspirin
* Active testicular or prostate cancer

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Total Score on the International Index of Erectile Function - Erectile Function | 6 week
  The International Index of Erectile Function - Erectile Function ( domain score is a patient questionnaire (six questions) used to measure various aspects of erectile performance and assess disease severity in efficacy trials concerning ED. The International Index of Erectile Function - Erectile Function has a minimum score of 0 and max of 30, higher scores mean a better outcome

SECONDARY OUTCOMES:
Total Erection Hardness Score | 6 week
  The Erection Hardness Score is a single-item scale that has demonstrated good psychometric properties for assessing erectile function in patients. The EHS has desirable measurement properties, including being highly responsive to treatment. This one-item PRO is robust and easy to use for evaluating erection hardness. The Total Erection Hardness Score has a minimum possible score of 0 and max of 4, higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Ranjodh S. Gill, MD, FACP, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No